CLINICAL TRIAL: NCT06251635
Title: Effects of Antipsychotics on Brain Insulin Action in Females: A Randomised Placebo-Controlled, Crossover Multi-Modal Neuroimaging Study
Brief Title: Effects of Antipsychotics on Brain Insulin Action in Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 127/2023
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Insulin Resistance; Menstrual Cycle; Type 2 Diabetes; Antipsychotics
Keywords: Antipsychotics; Brain Insulin Resistance; Magnetic Resonance Imaging (MRI); Metabolic Disturbances; Menstrual Cycle; Hyperinsulinemia; Insulin Lispro; Olanzapine; Physiological Effects of Drugs
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Hyperinsulinism | interventions — Olanzapine; Tablets; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study will follow a single-blind, crossover design wherein each participant will complete an MRI based protocol of brain insulin action. Participants will take part in two research visits during the follicular phase of their menstrual cycle (i.e., between day 4-10 of their menstrual cycle) and two visits during the luteal phase (between day 16-22, or within 5 days of next expected menses depending on individual cycle duration). In each cycle phase, participants will be given two doses of either oral olanzapine or oral placebo. After an overnight fast, fasting bloodwork will be obtained, followed by two MRI scans: one with intranasal placebo and one with intranasal insulin challenge (160 IU; 80 IU per nostril). Between scans they will have a short break and be asked to complete cognitive assessments/questionnaires.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to:
  1. Knowing whether they were assigned to the olanzapine or placebo conditions
  2. Knowing the order of the intranasal spray condition (insulin or placebo).
  Investigators will know when participants receive oral olanzapine or placebo and intranasal insulin or saline (required in order to schedule study assessments, and given the order of assessments on the MRI day). A separate staff member who is unaware of drug condition will administer cognitive assessments to mitigate bias of these outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follicular Phase Visits (Experimental): Participants will undergo two visits during the follicular phase of the menstrual cycle (they will be scanned between day 4-10 of their menstrual cycle). Each of the study periods will involve administration of OLA 5 mg HS (or PL) on day 0, OLA 10 mg HS (or PL) on day 1, and cognitive testing and MRI scanning on day 2. MRI assessments will occur 15 minutes after administering 160 International Units (IU) INI/INP.
  Interventions: Drug: Olanzapine 2.5Mg Oral Tablet; Drug: Placebo; Drug: Insulin Lispro 100 UNT/ML; Drug: Saline
- Luteal Phase Visits (Experimental): Participants will undergo two visits during the luteal phase of the menstrual cycle (they will be scanned between day 16-22, or within 5 days of next expected menses depending on individual cycle duration). Each of the study periods will involve administration of OLA 5 mg HS (or PL) on day 0, OLA 10 mg HS (or PL) on day 1, and cognitive testing and MRI scanning on day 2. MRI assessments will occur 15 minutes after administering 160 International Units (IU) INI/INP.
  Interventions: Drug: Olanzapine 2.5Mg Oral Tablet; Drug: Placebo; Drug: Insulin Lispro 100 UNT/ML; Drug: Saline

INTERVENTIONS:
Drug: Olanzapine 2.5Mg Oral Tablet — Olanzapine capsules (2.5mg) will be administered during one research visit for each menstrual cycle phase. The dosing schedule is as follows:
  1. Day 0- 5mg
  2. Day 1- 10mg
  Other Names: Apo-Olanzapine
Drug: Placebo — Placebo capsules visually identical to those containing olanzapine will be administered according to the same dosing schedule during one research visit of each menstrual cycle phase.
  Other Names: Olanzapine Placebo
Drug: Insulin Lispro 100 UNT/ML — At each visit, participants will be given an intranasal insulin challenge (160 IU) to assess brain insulin signalling via MRI based assay.
  Other Names: Intranasal Insulin
Drug: Saline — At each visit, participants will be given an intranasal saline placebo (1.6 mL) in order to establish baseline brain insulin signalling via MRI based assay.
  Other Names: Intranasal Saline

SUMMARY:
Females treated with antipsychotics have higher rates of comorbid metabolic syndrome than males. Despite this, females have historically been excluded from many mechanistic studies due to confounding effects of menstrual cycles. Recent evidence suggests that brain insulin resistance may be an underlying mechanism through which antipsychotics may exert their metabolic side effects. This study seeks to investigate how brain insulin action differs in females according to their menstrual cycle phase, and how a high metabolic liability agent such as olanzapine might interrupt these differential insulin effects. Young healthy females will be given olanzapine and intranasal insulin to test how these treatment combinations change brain processes. Participants will be tested during both the first half of their menstrual cycle (follicular phase) and the second half of their cycle (luteal phase). The investigators predict that intranasal insulin will change MRI-based measures in females, in a comparable way to males, in the follicular phase only. Adding olanzapine will block these effects of insulin in females in the follicular phase. This investigation has the potential to generate new knowledge in an area of significant unmet need. Demonstrating that antipsychotics disrupt brain insulin action, evidenced by inhibition of recognized effects of insulin on neuroimaging measures, will provide novel insights into currently poorly understood mechanisms.

DETAILED DESCRIPTION:
BACKGROUND: Antipsychotics (APs) cause serious metabolic adverse effects, including weight gain and type 2 diabetes. Females are disproportionally more affected by this problem than males. While the pathophysiology of these effects remain unclear, brain insulin resistance (IR) is posited to be an important determinant. Currently there are no direct methods to investigate brain IR, but physiological response to intranasal insulin (INI) can be used as a surrogate marker. INI reliably suppresses endogenous glucose production, modulates brain activity, and improves cognition. In a proof-of-concept neuroimaging study at CAMH, the investigators investigated AP-induced brain IR using an INI challenge. As expected, preliminary data show acute olanzapine (OLA) administration attenuates INI-induced changes in cerebral blood flow and resting state activity; however, the findings are only observed in males. It was recently suggested that brain insulin action differs between sexes, and this may relate to menstrual phases. Specifically, IR is physiologically induced in the luteal, but not follicular phase of the menstrual cycle. Hence, this study seeks to explore if the effects of APs on brain insulin action in females is modulated by menstrual stages.

HYPOTHESES: 1) INI, but not intranasal placebo (INP) will modulate resting state activity in the brain in females during the follicular phase of their menstrual cycle but not the luteal phase; 2) oral OLA will inhibit all INI-induced effects, relative to oral PL, during the follicular phase. OLA will have no apparent effect on females in the luteal phase given pre-existing brain IR.

APPROACH AND METHODOLOGY: Fifteen healthy normal weight (BMI <25 kg/m2), normal cycling female volunteers between the ages of 18-35 years will be recruited to participate in the study. In a single blind, crossover design, each participant will receive 4 treatment conditions (INP/PL, INI/PL, INP/OLA or INI-OLA) twice on 4 separate occasions (two visits per cycle phase). Each of the study periods will involve administration of OLA 5 mg HS (or PL) on day 0, OLA 10 mg HS (or PL) on day 1, and cognitive testing and MRI scanning on day 2. On Day 2, fasting blood work (glucose, insulin, c-peptide, olanzapine measures) will be followed by an MRI-based protocol of brain insulin action. This includes two MRI scans; one with intranasal insulin challenge (160 IU) and one with intranasal placebo. Study visits will take place 2-6 weeks apart to ensure specific menstrual phase across the four visits. Participants will undergo two visits during the follicular phase of the menstrual cycle (they will be scanned between day 4-10 of their menstrual cycle), and another two visits during the luteal phase of their menstrual cycle (between day 16-22, or within 5 days of next expected menses depending on individual cycle duration). Menstrual cycles will be tracked by self-report of the last three menstruation onset dates. Average cycle duration will be calculated to determine cycle phases. Based on this, participants will be invited to complete the visits during the specific windows of their follicular and luteal phase; measurement of sex hormones (progesterone, estrogen, luteinizing hormone (LH) and follicular stimulating hormone (FSH)) will be done at each visit to confirm cycle phase.

SIGNIFICANCE: Females suffer the most from AP-related metabolic adverse effects. Brain insulin action is increasingly being recognized as a potential mediator of these side effects. Disappointingly, females are an underrepresented population in the field because of the complex confounding effects of monthly hormonal variations. This is the first study to explore the effect of menstrual cycle phases on the anti-insulin action of APs. Thus, this investigation has the potential to generate new knowledge in an area of significant unmet need. Demonstrating that APs disrupt brain insulin action, evidenced by inhibition of recognized effects of INI on neuroimaging measures, will provide novel insights into currently poorly understood mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years
* Body Mass Index (BMI) between 18.5 - 24.9 kg/m2
* Normal menstrual cycle (defined as cycle length ranging from 21 to 35 days over the past 6 months).

Exclusion Criteria:

* History of psychiatric illness (screened using the Mini International Neuropsychiatric Interview (MINI));
* Pre-diabetes or diabetes (fasting glucose ≥6.0 mmol/L, HbA1c>6% or use of anti-diabetic drug);
* Evidence of impaired insulin sensitivity, assessed using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) ≥2.5;
* Family history of diabetes in a first degree relative (parent or sibling)
* Use of weight reducing agents;
* History of kidney or liver disease;
* Moderate-to-severe substance use;
* Irregular menstrual cycles (e.g., menstruation occurs less than 21 days or more than 35 days apart, or not having menstruated for three months (or 90 days), or conditions such as endometriosis or polycystic ovary syndrome (PCOS) or prior surgical interventions such as a hysterectomy or oophorectomy);
* Current use of hormonal birth control (e.g., pill, patch, hormonal intrauterine device [IUD], ring). Participants must have had at least 2 regular menstrual cycles following the discontinuation of hormonal birth control;
* Pregnant, gave birth in the last year, or breastfeeding. Participants must have at least 3 regular menstrual cycles post-breastfeeding before beginning the study;
* Current use of progesterone, estrogen, testosterone, or fertility treatment;
* Major medical or surgical event within the last 6 months;
* Any condition that interferes with safe acquisition of MRI data such as metal implants, pacemakers, cochlear implants, claustrophobia, etc.
* Any contraindications to the investigational products as listed in the product monographs including known hypersensitivity to the drug or the excipients of the product (note: enzymatic lactose intolerance is NOT exclusionary)
* Use of any of the prohibited medications listed in the product monograph of olanzapine (e.g., Levodopa and dopamine agonists and antihypertensive agents).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Resting State Functional Connectivity (assessed through Functional MRI) | Visits 1-4 (5-6 months); 2 visits during follicular phase, 2 visits during luteal phase. At each visit, either oral olanzapine or placebo is given. MRI #1 occurs after intranasal challenge #1 and MRI #2 occurs after intranasal challenge #2.
  Participants will complete 4 MRI scans to assess changes in resting state functional connectivity and activity across menstrual cycle phases and randomization conditions.Changes in resting state functional connectivity following intranasal insulin or placebo challenges, compared between the follicular and luteal phases of the menstrual cycle.

SECONDARY OUTCOMES:
Visuospatial Memory | Visits 1-4 (5-6 months) during break between MRI scan #1 and #2.
  Participants will complete the Brief Visuospatial Memory Test (BVMT) to assess visuospatial memory outcomes across the randomization conditions.
  BVMT Scoring: 0-36 (minimum 0, maximum 36)
Processing Speed | Visits 1-4 (5-6 months) during break between MRI scan #1 and #2.
  Participants will complete the Digit-Symbol Substitution Test (DSST) to assess processing speed across the randomization conditions.
  DSST Scoring: 0-110 (minimum 0, maximum 110)

CONTACTS AND LOCATIONS:
Overall Officials: Mahavir Agarwal, MBBS, PhD, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No